CLINICAL TRIAL: NCT07009392
Title: Microbiological Molecular Profile of the Knee Joint During Primary Reconstruction or Revision Surgery of the ACL
Acronym: INFECTIOGEN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2025-A00235-44
Record Dates: First submitted 2025-05-29; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: ACL - Anterior Cruciate Ligament Rupture
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NGS arm (Experimental)
  Interventions: Diagnostic Test: NGS Analysis

INTERVENTIONS:
Diagnostic Test: NGS Analysis — NGS (Next Generation Sequencing) analysis is performed on tissue from ACL

SUMMARY:
Anterior cruciate ligament (ACL) reconstructions are common surgical procedures, but a significant number fail for reasons that are not fully understood.

Silent infections have been shown to cause failure after other orthopedic surgical procedures such as fracture fixation and joint replacement. Silent and subclinical infections, as well as disruptions in the knee joint microbiome, could therefore be potential causes of failure after ligament reconstruction.

Traditional infection diagnostic methods (microbiological cultures) are often inadequate to detect these silent infections due to a lack of sensitivity. New molecular techniques such as high-throughput sequencing or NGS (next-generation sequencing) overcome this sensitivity problem and have proven effective in diagnosing polymicrobial infections.

Increased sensitivity compared to traditional culture has been reported in numerous studies, with some demonstrating the ability of NGS to isolate the infectious organism(s) in up to 82% of culture-negative cases.

These studies demonstrate the importance of advanced sequencing technologies for the diagnosis and management of infections after ACL reconstruction, offering promising prospects for improving clinical outcomes.

At the Jean Mermoz Private Hospital, ACL reconstruction is performed using a graft that is previously immersed in vancomycin. In this context, this study will characterize the knee joint microbiome in the context of ACL reconstruction with a graft treated with antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing primary ACL reconstruction or revision surgery
* Patient for whom access to the operative report of the primary ACL reconstruction is available
* Patient affiliated with or beneficiary of a social security system
* Patient who speaks French and has signed informed consent

Exclusion Criteria:

* Patients with preoperative signs or a history of knee joint infection
* Patients suffering from diabetes, cancer, or a chronic inflammatory disease
* Patients receiving immunosuppressive therapy
* Patients with elevated serum inflammatory markers
* Patients who have used intravenous drugs in the 3 months prior to surgery
* Patients who have used antibiotics in the 3 months prior to surgery
* Protected patients: adults under guardianship, curatorship, or other legal protection, persons deprived of their liberty by a judicial or administrative decision, persons under a protective measure, persons admitted to a health or social care facility for purposes other than research, and persons unable to express consent
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Knee microbiome description | Day 1
  Presence/absence of bacteria in knee joint of patients with ACL reconstruction

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé Jean Mermoz, Lyon, France